CLINICAL TRIAL: NCT02991677
Title: Exercise Effect on Chemotherapy-Induced Neuropathic Pain, Peripheral Nerve Fibers
Brief Title: Exercise Effect on Chemotherapy-Induced Neuropathic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alice S. Ryan, PhD, Professor, Baltimore VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00070946
Record Dates: First submitted 2016-11-30; First posted 2016-12-13 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cancer, Breast; Cancer, Colorectal; Cancer, Lung; Cancer, Ovarian
Keywords: exercise; neuropathy
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Other): This is an attention control group with regular contact by study staff.
  Interventions: Other: control group
- aerobic exercise (Experimental): Aerobic exercise intervention is for 12 weeks 3 times weekly with training on site.
  Interventions: Behavioral: aerobic exercise intervention
- resistive training (Experimental): Intervention is for 12 weeks 3 times weekly with training on site.
  Interventions: Behavioral: resistive training

INTERVENTIONS:
Behavioral: aerobic exercise intervention — Exercise physiologist supervised walking or running on the treadmill 3 times weekly for 12 weeks.
  Arms: aerobic exercise
Other: control group — weekly contact by study staff with survivorship information offered not related to neuropathy.
  Arms: control
Behavioral: resistive training — Exercise physiologist supervised upper and lower extremity resistive training 3 times weekly for 12 weeks
  Arms: resistive training

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) continues to be a serious healthcare concern. It is painful, persistent, resistant to conventional pain therapies, and results in long-term suffering and decreased quality of life for many cancer survivors. The role of exercise to decrease CIPN-related neuropathic pain (CIPN-NP) will be investigated, with the goal of identifying the mechanisms associated with this therapeutic approach to manage CIPN-NP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with cancer, stage I-IV
* History of treatment with oxaliplatin, docetaxel, or paclitaxel, either alone or in combination with other agents
* Completion of chemotherapy > 6 months < 1 year
* Ability to walk on a treadmill
* Medical clearance from oncologist or primary care provider
* Presence of CIPN per National Cancer Institute Common Toxicity Criteria grade 1-3 (0-no signs/symptoms, 1-minor loss of function, 2-increased symptoms not interfering with activities of daily living (ADLs), 3-severe symptoms interfering with ADL, 4-disabling, and 5 is death)
* Score on Neuropathic Pain Scale >1
* Age 21-70

Exclusion Criteria:

* Denial of CIPN
* Other motor/sensory neuropathy caused by other than chemotherapy (i.e.alcohol-related, autoimmune diseases, diabetes)
* Coronary artery disease
* History of >1 chemotherapy regimen
* Musculoskeletal conditions which preclude participation in an exercise training program
* Pregnancy
* Regular exerciser, defined as >90 minutes per week of aerobic exercise and any resistive training

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensory pain | 13 weeks
  Thermal, mechanical, and vibration sensation by quantitative sensory testing

SECONDARY OUTCOMES:
Nerve fiber density | 13 weeks
  laboratory examination of skin biopsy samples for measurement of nerve fiber density

CONTACTS AND LOCATIONS:
Overall Officials: Alice Ryan, PhD, Principal Investigator — University of Maryland at Baltimore School of Medicine
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided